CLINICAL TRIAL: NCT03743831
Title: Comparison of Haemodynamic Effects During Orotracheal Intubation, by Direct or Indirect Laryngoscopy With Airtraq, Controlled, Prospective, Randomized, Simple-blind, Monocentric Study at the Lille University Hospital Specialties Block.
Brief Title: Comparison of Haemodynamic Effects During Orotracheal Intubation, by Direct or Indirect Laryngoscopy With Airtraq
Acronym: HEMODAIRTRAQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Vygon GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2017_72; 2018-A01683-52 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Orotracheal Intubation
Keywords: Laryngoscopy direct; Laryngoscopy indirect by Airtraq; hemodynamic changes; side effects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- orotracheal intubation direct (Other)
  Interventions: Device: orotracheal intubation by direct laryngoscopy
- orotracheal intubation indirect (Other)
  Interventions: Device: orotracheal intubation by indirect laryngoscopy

INTERVENTIONS:
Device: orotracheal intubation by direct laryngoscopy — Orotracheal intubation by direct laryngoscopy by metal blade type Macintosch
  Arms: orotracheal intubation direct
Device: orotracheal intubation by indirect laryngoscopy — orotracheal intubation by indirect laryngoscopy by Airtraq
  Arms: orotracheal intubation indirect

SUMMARY:
News techniques of intubation by indirect laryngoscopy have arrived in operating rooms but they are still too restricted to situations (difficult intubation criteria ..). It wanted to focus on indirect laryngoscopy by Airtraq. This technique allows better exposure during intubation while limiting mouth opening and cervical hyper extension, but also dental trauma and lip wounds. It also reduces the duration of laryngoscopy and therefore at the same time the apnea time. After a review of the literature, it has been proven that its use reduces haemodynamic changes during intubation. But these studies have been realized only in very particular patients (obese, heart failure) and with induction protocols that are not used routinely in our operating theaters.

Reasons why it decided to carry out this study, on the one hand to find these results and especially to be able to extend them to the whole population.

ELIGIBILITY:
Inclusion Criteria:

* Specific medical conditions: ASA 1 or 2
* Patient having given written consent to participate in the category 2 trial
* Intubation realized by experienced person
* Social Insured Patient
* Patient willing to comply with all procedures of the study and its duration

Exclusion Criteria:

* Demographic characteristics: minor, over 65
* Medical history: history of difficult intubation, hypertension
* Lille intubation score greater than or equal to 7
* Treatments in progress: Beta taking blocking the day of the operation.
* Administrative reasons: inability to receive informed information, inability to participate in the entire study, lack of coverage by the social security system, refusal to sign consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
change from intubation mean blood pressure at 1 min after intubation | between the values before intubation (T0) and 1min after intubation.

SECONDARY OUTCOMES:
Frequency of patients with hemodynamic reaction post intubation (minimal variation of mean blood pressure or heart rate of 20% | between values before intubation and 1, 2, 5, 10 minutes after intubation.
Variation of blood pressure (PAM) | between the values before intubation (T0) and 2, 5 and 10 minutes of intubation
Variation of heart rate (HR) | between the values before intubation (T0) and 1, 2, 5 and 10 minutes of intubation
Mean of the arterial blood pressure and heart rate | before intubation and at 1,2,5 and 10 minutes from intubation.
  delta defined by the difference between the values
Intubation time in seconds from introduction of the intubation device into the mouth with inflation of the balloon | at 1 min after intubation
Frequency of patients with dental trauma and / or an injury to the lips due to the intubation device. | at 10 min after intubation
instantaneous ANI delta | between ANI before intubation and 1,2,5 and 10 min after intubation

CONTACTS AND LOCATIONS:
Overall Officials: Elsa Jozefowicz, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France